CLINICAL TRIAL: NCT01138358
Title: Experiences of Episodic Breathlessness (EB) in Patients With Advanced Disease
Brief Title: Study of Episodic Breathlessness in Patients With Lung Cancer or Other Advanced Disease
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000674580; UKM-KCH-EB-V4; EU-21039
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-06

CONDITIONS: Dyspnea; Lung Cancer; Metastatic Cancer
Keywords: dyspnea; lung metastases; recurrent non-small cell lung cancer; recurrent small cell lung cancer; extensive stage small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Dyspnea; Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

INTERVENTIONS:
Other: medical chart review
Other: study of socioeconomic and demographic variables
Other: survey administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about experiences of episodic breathlessness in patients with advanced disease may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying experiences of episodic breathlessness in patients with lung cancer or other advanced disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To explore the experiences of episodic breathlessness in patients with advanced disease (i.e., primary and secondary lung cancer, chronic obstructive pulmonary disease [COPD], chronic heart failure [CHF], and motor neuron disease [MND]).
* To explore the impact of episodic breathlessness on daily living.
* To explore the individual coping strategies to reduce burden of episodic breathlessness.

OUTLINE: This is a multicenter study.

Patients undergo 1 to 2 interviews to collect data on experiences of breathlessness (in general, at rest, and on exertion including symptom description, interpretation, and meaning); experiences of episodic breathlessness (EB) (at rest and on exertion including symptom description, interpretation, meaning, and definition); trajectory/course of EB (onset/relief, time, and severity) and different types/trajectories of EB; impact of EB (burden, emotional reaction [panic and fear], care burden, and dependencies); triggers of EB (causes, situation, and settings) and predictability of EB; management of EB (coping strategies, non-pharmacological and pharmacological management [including different applications], worsen/relief, role of care in coping, and emotional/behavior strategies; views on and experiences with services/professionals in management of EB and response to professional advice; and attitudes towards the future, course of the disease, and awareness of prognosis. At the end of the interview, the patient will be asked to draw a figure that illustrates the trajectory of the episode. After the interview, a debriefing will be carried out to give the patient the chance to express worries, potential harm, or any comments about the interview. In addition to the interviews, further information will be collected including demographics, diagnosis and co-morbidities, current pharmacological and non-pharmacological treatments (medical history), functional status (Karnofsky), and breathlessness characteristics (e.g., intensity, frequency, and duration). The interviews will be tape-recorded, transcribed verbatim, and analyzed concurrently using Framework Approach.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced disease as defined by the following criteria:

  * Lung cancer

    * Primary lung cancer at all stages (small cell lung cancer [SCLC] and non-small cell lung cancer [NSCLC])
    * Cancer at any site with secondary tumor of the lung (lung metastasis)
  * Chronic obstructive pulmonary disease (COPD)

    * Stage III or IV of the Global Initiative for Obstructive Lung Disease (GOLD) classification, which includes the airflow limitation measured by spirometry FEV1 < 50%, FEV1/FVC < 0.7, and symptoms such as more severe breathlessness, reduced exercise capacity, and repeated exacerbations
  * Chronic heart failure (CHF)

    * NYHA class II-IV heart disease, which includes symptoms such as dyspnea or palpitation and an increasing limitation of exercise capacity or discomfort at rest
  * Motor neuron disease (MND)

    * All patients suffering from breathlessness
* Suffering from episodic breathlessness as defined above at any level of severity

PATIENT CHARACTERISTICS:

* Able to give informed consent
* Able to be interviewed
* No cognitive impairment (clinically judged by the principal investigator)
* No limited comprehension of the English language

PRIOR CONCURRENT THERAPY:

* Concurrent disease-oriented therapies (e.g., chemotherapy, radiotherapy, or surgery) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Experiences of episodic breathlessness
Impact of episodic breathlessness on daily living
Individual coping strategies to reduce burden of episodic breathlessness

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Simon, MD, MSC, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, England, United Kingdom

REFERENCES:
- [Derived] Simon ST, Niemand AM, Benalia H, Voltz R, Higginson IJ, Bausewein C. Acceptability and preferences of six different routes of drug application for acute breathlessness: a comparison study between the United Kingdom and Germany. J Palliat Med. 2012 Dec;15(12):1374-81. doi: 10.1089/jpm.2012.0249. Epub 2012 Oct 24. PMID 23094954